CLINICAL TRIAL: NCT06665243
Title: Effects of Technology-Enhanced Horticultural Activities Among the People with Dementia and Their Family Caregivers
Brief Title: Horticultural Activities Among the People with Dementia and Their Family Caregivers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Patrick KOR Pui Kin, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBA20241029
Record Dates: First submitted 2024-10-28; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Dementia; Caregiver Stress
Keywords: horticultural therapy; horticultural activities; people with dementia; family caregivers; informal caregivers; technology-enhanced horticultural activities
MeSH Terms: conditions — Dementia; Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Technology-enhanced horticultural activities (Experimental)
  Interventions: Behavioral: Technology-enhanced horticultural activities

INTERVENTIONS:
Behavioral: Technology-enhanced horticultural activities — The indoor technology-enhanced horticultural activities will be delivered to people with dementia and their family caregivers through a smart grower. The smart grower is a hydroponic indoor grower that creates a controllable environment with auto optimization for growing healthy plants, fresh vegetables, herbs, and fruits. A mobile app will be connected to the grower for controlling the growing environment (e.g., lighting, watering), tracking the progress of the plants, and guiding the older people with dementia and their family caregivers in conducting the horticultural activities. The program will consist of eight face-to-face (F-T-F) horticultural activity training sessions for groups of 6-8 participants. The indoor program contains various horticultural, cognitive, and multisensory stimulation activities, such as asking PWD and family caregivers to record the sense of touch and odor when caring for the plants and to observe the various changes in the plants using the smart grower.

SUMMARY:
The goal of this study is to explore the effects of technology-enhanced horticultural activities on people with dementia (PWD) and their family caregivers. The main questions it aims to answer are:

* Do these activities improve cognitive function and behavioral symptoms in PWD?
* Do they reduce stress and depressive symptoms in caregivers and improve their quality of life?

The study will have two phases:

* Phase I: Conduct a pilot study with PWD in a geriatric day hospital to evaluate feasibility and initial effects.
* Phase II: Conduct a larger trial with PWD and caregivers in community settings to further assess impact.

Participants will engage in indoor horticultural activities using a smart grower, participate in training sessions, and complete assessments before and after the intervention.

DETAILED DESCRIPTION:
Dementia is becoming a major worldwide concern as the world's population ages and the prevalence of dementia increases exponentially with age. As the disease progresses, people with dementia (PWD) exhibit different behavioral symptoms, and their cognitive function and self-care ability gradually decline. The burden of caring and the uncertainty about disease progression result in high levels of stress and negative emotions in family caregivers.

Horticultural therapy is an effective intervention that has been shown to increase the time PWD spend engaging in leisure activities and decrease the time they spend doing nothing. Importantly, horticultural therapy has demonstrated positive effects on alleviating agitation behaviors among PWD, including harmful aggressive and destructive behaviors. PWD can also benefit from improved cognitive function, psychological symptoms (e.g., stress, depression), and enhanced social interaction when participating in horticultural therapy.

However, there are limitations and constraints for PWD to participate in horticultural therapy, especially in high-density cities like Hong Kong. First, the majority of PWD and their family caregivers cannot afford to have a garden within their homes, as many developed cities suffer from limited land space, and it is common for PWD and their caregivers to live in small areas with simple furniture. Second, uncontrollable weather contributes to the difficulty in performing horticultural therapy in outdoor conditions, as plants are sensitive to weather and vulnerable to unstable conditions, especially the fickle weather in Hong Kong. Third, insufficient human resources lead to an increased chance of failure in outdoor horticultural therapy, as it requires ample manpower to look after the condition of various plants and assist PWD and their caregivers during the therapy sessions. Therefore, performing indoor technology-enhanced horticultural activities with a smart grower machine has the potential to reduce concerns about space, weather, and manpower.

The study consists of two phases. Phase I is a pilot pre-post feasibility study conducted in a geriatric day hospital setting with 30 PWD participants. It aims to assess whether indoor technology-enhanced horticultural activities improve cognitive function and behavioral symptoms in PWD. Phase II involves a larger-scale single-arm trial with 100 pairs of PWD and caregivers in community settings to evaluate the dyadic approach's impact on caregivers' stress levels and quality of life.

The intervention uses a smart grower, an indoor hydroponic system, to facilitate horticultural activities. A mobile app assists in controlling the environment and guiding participants. The program includes eight face-to-face sessions with various cognitive and sensory activities.

Primary outcomes for PWD include engagement, cognitive functioning, and challenging behaviors. Caregivers' outcomes focus on positive caregiving experiences, perceived stress, quality of life, and depressive symptoms. Feasibility is assessed through recruitment, attendance, completion, and retention rates. Evaluations will be conducted at baseline (0 weeks) and post-intervention (8 weeks).

ELIGIBILITY:
Inclusion Criteria (PWD):

* aged 65 or above;
* diagnosed with any type of dementia at the early to moderate stage;
* community-dwelling (i.e., non-institutionalized); and
* able to understand Cantonese and follow simple instructions.

Inclusion Criteria (Caregivers)

* aged 18 years or above;
* blood or by-marriage relatives (e.g., spouses, siblings, children, and grandchildren) of a person who has been clinically diagnosed with dementia, regardless of its type;
* are taking up caring responsibilities ranging from physical aid to emotional support, in the form of transportation, financial assistance, personal hygiene, and decision-making;
* providing most of the daily care and support for PWD (daily contact for at least four hours); and
* able to speak Cantonese.

Exclusion Criteria (PWD + Caregivers):

* being diagnosed with a mental disorder such as bipolar disorder, schizophrenia, or depression;
* taking anticonvulsants or any kind of psychotropic drugs; and
* identified with self-reported suicidal thoughts or drug abuse in the past 6 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
PWD Outcome: Cognitive Functioning | 8 Weeks
  The MoCA-5-min will assess participants' cognitive function (Wong et al., 2015). It covers four domains: attention, executive function/language, orientation, and memory. The MoCA-5-min is highly correlated with the MoCA (r = 0.87) and has excellent test-retest reliability (ICC = 0.89). Trained nursing students will conduct the MoCA-5-min assessments.
PWD Outcome: Engagement | 8 Weeks
  The Engagement of a Person with Dementia Scale (EPWDS) assesses behavioral and emotional engagement in individuals with dementia during psychosocial activities (Jones et al., 2018). Based on the Observational Method of Engagement (Cohen-Mansfield et al., 2009), it evaluates five areas: affective, visual, verbal, behavioral, and social engagement. Each area includes two items-one for positive engagement and one for disengagement-resulting in 10 items total. Negatively phrased items are reverse scored, with total scores ranging from 10 to 50, where higher scores indicate greater positive engagement. The EPWDS has excellent reliability, with an internal consistency of 0.94 and a test-retest reliability of r = 0.95 (Jones et al., 2018).
  In this study, two trained nursing students will administer the EPWDS through direct observations and field notes. Inter-rater reliability will be calculated to ensure consistent assessments. Observations will last for 10 minutes and occur at T0 and T1.
PWD Outcome: Challenging Behaviors | 8 Weeks
  The Challenging Behaviors Subscale of the Dementia Coding System (DeCS) will measure challenging behaviors in BPSD during the intervention (Hillebrand et al., 2023). The DeCS uses a systematic time-sampling approach, observing individuals with dementia at specific intervals. The subscale includes 18 behaviors (e.g., apathetic, tense posture, runs away) recorded on a dichotomous scale, where 0 indicates not observed and 1 indicates observed. A higher score indicates more challenging behaviors. The subscale's internal consistency is 0.71, and the test-retest reliability is ICC = 0.92 (Hillebrand et al., 2023). Two trained nursing students will conduct observations and take field notes using the DeCS. Inter-rater reliability will be calculated to ensure consistency. Observations will be conducted over five four-minute intervals at T0 and T1.
PWD Outcome: Challenging Behaviors | 8 Weeks
  Challenging behaviors of the PWD will be measured by the Chinese version of the Neuropsychiatric Inventory-Questionnaire (NPI-Q) (Wong et al., 2014), administered by caregivers. It evaluates the frequency, severity, and caregiver distress of 12 neuropsychiatric symptoms using a 5-point rating scale. The NPI-Q has acceptable psychometric properties, including a high internal consistency (α = 0.76) and test-retest reliability (0.99).
Caregivers' Outcome: Positive Caregiving Experience | 8 Weeks
  The Chinese version of the Positive Aspect of Caregiving scale (PAC) (Lou et al., 2015) will measure participants' positive caregiving experience. The PAC scale demonstrates acceptable internal consistency (α = 0.85) among family caregivers of PWD in Hong Kong. Higher scores indicate more positive self-perceptions of caregiving.
Caregivers' Outcome: Perceived Stress Level | 8 Weeks
  The Chinese version of the Perceived Stress Scale (PSS) will measure participants' perceived stress (Leung et al., 2010). The PSS contains 10 items rated on a 5-point Likert scale from 0 (never) to 4 (very often). It has acceptable psychometric properties, including internal consistency (α = 0.85) and test-retest reliability (0.85) (Chu & Kao, 2005; Leung et al., 2010).
Caregivers' Outcome: Quality of Life | 8 Weeks
  The WHOQOL-OLD BREF (HK) will assess participants' quality of life (QOL) (Leung et al., 2005). It comprises 28 items, each rated on a 5-point Likert scale from 1 (very dissatisfied) to 5 (very satisfied), with higher scores indicating better QOL. The internal consistency of the Hong Kong Chinese version of the WHOQOL is satisfactory, with Cronbach's alpha ranging from 0.73 in the environment domain to 0.83 in the psychological domain, and a test-retest reliability coefficient of 0.83.
Caregivers' Outcomes: Depressive Symptoms | 8 Weeks
  The Chinese version of the Center for Epidemiological Studies Depression scale (CESDS) (Chin et al., 2015) will measure depression. It is a self-reported measure containing 20 items (Radloff, 1977). The CESD has acceptable psychometric properties, including test-retest reliability (0.91) and internal consistency for general depression (α = 0.86).

SECONDARY OUTCOMES:
Feasibility Outcome: Recruitment Rate | 8 Weeks
  The ratio of participants enrolled to the total number approached.
Feasibility Outcome: Attendance Rate | 8 Weeks
  The average number of sessions attended by participants relative to the total sessions offered.
Feasibility Outcome: Completion Rate | 8 Weeks
  The proportion of participants who complete at least 80% of required assessments and interventions compared to those initially enrolled.
Feasibility Outcome: Retention Rate | 8 Weeks
  The percentage of participants who remain in the study from T0 through T1.

IPD SHARING:
Plan to Share IPD: No